CLINICAL TRIAL: NCT05650034
Title: Post-Operative Radiotherapy De-Escalation of Negative Nodal Regions in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO2105-30901
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Carcinoma
Keywords: Post operative radiotherapy; Elective nodal irradiation; Head and neck SCC; Elective nodal omission; De-escalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elective nodal de-escalation arm (Experimental): Omission of elective nodal irradiation in N0 hemi-neck of well lateralized H&N SCCs ( pN0 or by PETCT). Dose de-escalation of elective nodal irradiation in N0 hemi-neck of midline H&N SCCs ( pN0 or by PETCT).
  Interventions: Radiation: Elective nodal de-escalation arm

INTERVENTIONS:
Radiation: Elective nodal de-escalation arm — Omission of elective nodal irradiation in N0 hemi-neck of well lateralized H&N SCCs ( pN0 or by PETCT). Dose de-escalation of elective nodal irradiation in N0 hemi-neck of midline H&N SCCs ( pN0 or by PETCT).

SUMMARY:
This is a non-randomized prospective trial evaluating the non- inferiority of de-escalating the volume and/or dose of elective nodal irradiation in post-operative head and neck squamous cell carcinomas.

DETAILED DESCRIPTION:
This is a non-randomized prospective trial evaluating the non-inferiority of volume and/or dose de-escalation of elective nodal irradiation in post-operative head and neck squamous cell carcinomas with assessment of toxicity profiles.

57 head and neck squamous cell carcinoma cases eligible for post-operative radiotherapy will be recruited and managed according to tumor laterality, nodal status, and laterality of nodal dissection (ipsilateral/ bilateral nodal dissection).

Ipsilateral nodal dissection:

* If ipsilateral N0, bilateral nodal irradiation will be omitted.
* If ipsilateral N positive and tumor was well lateralized, contralateral nodal negativity will be assessed by PETCT. IF PETCT is free, the ipsilateral nodal regions will be irradiated with conventional doses while the contralateral nodal irradiation will be omitted.
* If ipsilateral N positive and tumor was not well lateralized, ipsilateral nodal regions will be irradiated with conventional doses while the contralateral nodal irradiation will be de-escalated to 40 Gy dose equivalent.
* Cases with PETCT positive for malignancy will be excluded from the study.

Bilateral nodal dissection:

* If bilateral N0, bilateral nodal irradiation will be omitted.
* If one sided N positive, laterality of the tumor will be assessed:

  * In well lateralized tumors, the positive side nodal regions will be irradiated while the contralateral nodal irradiation will be omitted.
  * In midline/ non lateralized tumor the positive side nodal regions will be irradiated with conventional doses while the contralateral nodal irradiation will be de-escalated to 40 Gy dose equivalent.
* If bilateral N positive, cases will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Karnofsky performance score of 70% or more.
* Completely or partially resected head and neck SCC. This includes: The oral cavity (lips, buccal mucosa, oral tongue, floor of mouth, gingiva, retromolar trigone, and hard palate), maxilla, oropharynx, and larynx.
* Patients with at least an ipsilateral neck dissection.
* Patient has at least one pathological feature that is an indication for PORT: positive or close (<5 mm) margin, presence of LVI or PNI, pT3 or pT4 disease, positive lymph nodes, or ENE.
* Pathologically lymph node negative in at least one dissected hemi-neck or PET-CT

Exclusion Criteria:

* Patients with bilaterally involved neck nodes
* Patients with pT3-T4 tumors involving midline who undergo an ipsilateral neck dissection (unless a contralateral neck dissection is performed)
* Serious medical comorbidities or other contraindications to radiotherapy
* Prior history of head and neck cancer within 5 years
* Any other active invasive malignancy
* Prior head and neck radiation at any time
* Prior oncologic head and neck surgery in the oral cavity or neck.
* Known metastatic disease
* Locoregional disease recurrence identified following surgical resection but prior to start of radiotherapy
* Inability to attend full course of radiotherapy or follow-up visits 11.Unable or unwilling to complete QoL questionnaires

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Regional failure in the omitted/de-escalated elective nodal irradiation site | Baseline to 1 year

SECONDARY OUTCOMES:
Acute toxicity | Baseline to 6 months
Late toxicity | Baseline to 1 year
Overall survival | Baseline to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shouman, Study Director — National Cancer Institute, Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided